CLINICAL TRIAL: NCT03062527
Title: Effects of Low and Versus Moderate Glycemic Index Diets on Physical Capacity and Body Composition in Endurance- Trained Runners
Brief Title: Effect of Glycemic Index on Physical Capacity in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, PhD, Assistant Professor, Poznan University of Life Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ULS00001
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Nutrition; Sport; Glycemic Index; Physical Capacity
Keywords: Nutrition; Training support; Low Glycemic Index; Moderate Glycemic Index; Endurance; Running

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Index Diet (Experimental): Group consuming low glycemic index diet. Calculated glycemic index of daily diet was lower than 40. Carbohydrate- containing foods included whole rye bread, pumpernickel bread, whole oats, wheat brans, brown rice, buckwheat, vegetables (besides corn, cooked carrots, potatoes and pumpkin) and fruit such as apples, pears, grapefruits, tangerines, prunes, dried apricots and unripe bananas.
  Interventions:
  The experimental procedure for each participant included a 3-week low glycemic index diet. Between the 3-week low and moderate glycemic index diets or a moderate and low glycemic index treatment, a 14-day washout period was introduced.
  Interventions: Other: Dietary Intervention: Low vs. moderate glycemic index
- Moderate Glycemic Index Diet (Experimental): Group consuming moderate glycemic index diet. Calculated glycemic index of diet was higher than 60. Carbohydrate- containing foods included wheat bread, wheat rolls, potatoes, instant oats, cornflakes, white rice, millet, boiled carrots and fruit (ripe bananas, grapes, raisins, dates, cranberry, honey and high sugar jams)
  Interventions:
  The experimental procedure for each participant included a 3-week moderate glycemic index diet. Between the 3-week low and moderate glycemic index diets or a moderate and low glycemic index treatment, a 14-day washout period was introduced.
  Interventions: Other: Dietary Intervention: Low vs. moderate glycemic index

INTERVENTIONS:
Other: Dietary Intervention: Low vs. moderate glycemic index

SUMMARY:
The purpose of the present study was to assess the influence of low vs moderate glycemic index of a 3-week diet on aerobic capacity, endurance performance and body mass and composition in endurance-trained athletes in a randomized, controlled crossover trial.

DETAILED DESCRIPTION:
The effect of glycemic index of pre-exercise meal on endurance capacity and performance has been widely investigated. However, little is known about the adaptations to longer dietary interventions with different glycemic index and their influence on aerobic capacity and body composition in runners. Therefore, the purpose of this study was the assessment of the influence of low GI vs moderate GI of a 3-week diet on aerobic capacity, endurance performance and body mass and composition in endurance-trained athletes in a randomised, controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* male and female,
* a current medical clearance to practice sports,
* training experience: at least 3 years,
* minimum of 4 workout sessions a week lasting at least 1.5-2 hours/day,
* age: 17 - 37 years.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol,
* smoking, illicit drug use, alcohol consumption greater than 1-2 drinks/week, dietary supplements use less than 3 weeks before the study,
* females- being pregnant or planning to become pregnant during the study.

Ages: 17 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-02-06 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in aerobic capacity following low glycemic index diet | Baseline and after 3 weeks
Changes in aerobic capacity following moderate glycemic index diet | Baseline and after 3 weeks
Changes in performance in 12-min running test following low glycemic index diet | Baseline and after 3 weeks
Changes in performance in 12-min running test following moderate glycemic index diet | Baseline and after 3 weeks
Changes in fat mass and fat free mass following low glycemic index diet | Baseline and after 3 weeks
  Fat mass (kg) and fat free mass (kg) analysis
Changes in fat mass and fat free mass following moderate glycemic index diet | Baseline and after 3 weeks
  Fat mass (kg) and fat free mass (kg) analysis

SECONDARY OUTCOMES:
Statistical evaluation of the significance of differences between the changes in aerobic capacity indices | 1 year
Statistical evaluation of the significance of differences between the changes in performance in 12-min running test | 1 year
Statistical evaluation of the significance of differences between the changes in fat mass and fat free mass | 1 year
  Fat mass (kg) and fat free mass (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jeszka, Professor, Study Chair — Department of Hygiene and Human Nutrition, Poznan University of Life Sciences, Poznan, Poland
Locations (1):
- Poznan University of Life Sciences, ul.Wojska Polskiego 31, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level recorded indicators (body composition, aerobic capacity, performance in 12-min running test), without personal data. Depending on the requirements of the journal, the data obtained will be attached to scientific publications, deposited in a public repository or provided by principal investigator when requested.